CLINICAL TRIAL: NCT02347605
Title: Medicinal Nicotine for Preventing Cue Induced Craving
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: WS2385492
Record Dates: First submitted 2015-01-14; First posted 2015-01-27 (Estimated); Results first posted 2017-12-18 (Actual); Last update posted 2017-12-18 (Actual); Status verified 2017-12

CONDITIONS: Tobacco Use Disorder
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Tobacco Use Cessation Devices

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Nicotine lozenge 4 mg prior to cue exposure (Experimental): Nicotine lozenge is used 15 minutes prior to smoking cue exposure
  Interventions: Drug: Nicotine lozenge 4 mg
- Placebo lozenge prior to cue exposure (Placebo Comparator): Placebo lozenge is used 15 minutes prior to smoking cue exposure
  Interventions: Drug: Placebo lozenge
- Control condition: Lozenge after cue exposure (Other): Lozenge is used immediately after smoking cue exposure
  Interventions: Drug: Nicotine lozenge 4 mg

INTERVENTIONS:
Drug: Nicotine lozenge 4 mg
  Arms: Control condition: Lozenge after cue exposure; Nicotine lozenge 4 mg prior to cue exposure
Drug: Placebo lozenge
  Arms: Placebo lozenge prior to cue exposure

SUMMARY:
The purpose of this study is to determine if changing the timeframe (relative to cue presentation) at which the nicotine lozenge is given can attenuate the increase in symptoms of tobacco craving and withdrawal that occur when smokers are presented with smoking cues. In this cross-over study, all subjects attend three laboratory sessions at which either nicotine lozenge or placebo is given prior to presentation of smoking cues or after presentation of smoking cues. The order in which the three conditions will be presented are randomized.

ELIGIBILITY:
Inclusion Criteria:

* Smoking a minimum number of cigarettes per day
* General good health

Exclusion Criteria:

* unstable medical or psychiatric conditions
* history of severe motion sickness (due to virtual reality equipment used to present cues)
* women who are pregnant or breast feeding

The investigators will evaluate if there are other reasons why someone may not participate

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2013-09; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Kotlyar, PharmD, Principal Investigator — University of Minnesota
Locations (1):
- Clinical and Translational Sciences Institute, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Sequence 1: Placebo lozenge 15 minute prior to cue exposure at lab 1; Nicotine lozenge 15 minutes prior to cue exposure at lab 2; Nicotine lozenge after cue exposure at lab 3
- Sequence 2: Placebo lozenge 15 minute prior to cue exposure at lab 1; Nicotine lozenge after cue exposure at lab 2; Nicotine lozenge 15 minutes prior to cue exposure at lab 3
- Sequence 3: Nicotine lozenge 15 minutes prior to cue exposure at lab 1; Placebo lozenge 15 minute prior to cue exposure at lab 2; Nicotine lozenge after cue exposure at lab 3
- Sequence 4: Nicotine lozenge 15 minutes prior to cue exposure at lab 1; Nicotine lozenge after cue exposure at lab 2; Placebo lozenge 15 minute prior to cue exposure at lab 3
- Sequence 5: Nicotine lozenge after cue exposure at lab 1; Placebo lozenge 15 minute prior to cue exposure at lab 2; Nicotine lozenge 15 minutes prior to cue exposure at lab 3
- Sequence 6: Nicotine lozenge after cue exposure at lab 1; Nicotine lozenge 15 minutes prior to cue exposure at lab 2; Placebo lozenge 15 minute prior to cue exposure at lab 3
Period: Overall Study
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6
Started | 10 | 10 | 8 | 10 | 9 | 9
Completed Lab 1 | 10 | 10 | 8 | 10 | 8 | 9
Completed Lab 2 | 7 | 7 | 7 | 7 | 6 | 8
Completed (Completed lab 3 (and therefore the entire study)) | 7 | 7 | 7 | 6 | 6 | 7
Not Completed | 3 | 3 | 1 | 4 | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6 | Total
Number analyzed (Participants) | 10 | 10 | 8 | 10 | 9 | 9 | 56
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.1 (12.1) | 45.9 (11.6) | 40.1 (16.6) | 37 (12.1) | 48.6 (12.3) | 48.7 (11.6) | 43.1 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 3 | 5 | 6 | 5 | 28
  Male | 6 | 5 | 5 | 5 | 3 | 4 | 28
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 0 | 1 | 2
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 7 | 1 | 0 | 4 | 3 | 3 | 18
  White | 3 | 8 | 7 | 3 | 6 | 5 | 32
  More than one race | 0 | 1 | 1 | 1 | 0 | 0 | 3
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 8 | 10 | 9 | 9 | 56

OUTCOME MEASURES:

1. Primary Outcome: Craving Symptom Severity Score Assessed Via Questionnaire
Description: Craving as assessed via the craving question on the Minnesota Nicotine Withdrawal Scale. The score range is from 0 (no craving) to 4 (severe craving). The outcome measure is the change in craving score from before cue exposure to craving score after cue exposure.
Time Frame: approximately 15 minutes
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Nicotine Lozenge Prior to Cue Exposure: Nicotine lozenge is used 15 minutes prior to smoking cue exposure
  Nicotine lozenge 4 mg
- Placebo Lozenge Prior to Cue Exposure: Placebo lozenge is used 15 minutes prior to smoking cue exposure
  Placebo lozenge
- Control Condition: Lozenge After Cue Exposure: Lozenge is used immediately after smoking cue exposure
  Nicotine lozenge 4 mg
Arm/Group | Nicotine Lozenge Prior to Cue Exposure | Placebo Lozenge Prior to Cue Exposure | Control Condition: Lozenge After Cue Exposure
Number analyzed (Participants) | 46 | 46 | 45
units on a scale | 0.52 (0.13) | 0.57 (0.13) | 0.31 (0.13)
Statistical Analysis 1: Comparison: Nicotine Lozenge Prior to Cue Exposure vs Placebo Lozenge Prior to Cue Exposure vs Control Condition: Lozenge After Cue Exposure; Test type: Superiority; p = 0.25, Mixed Models Analysis — Adjusted for treatment order, session, room sequence

2. Primary Outcome: Withdrawal Symptom Severity Score Assessed Via Questionnaire
Description: Withdrawal as assessed via the Minnesota Nicotine Withdrawal Scale. The score range is from 0 to 28 with higher scores indicating more severe withdrawal symptoms. The outcome measure is the change in withdrawal score from before cue exposure to the withdrawal score after cue exposure.
Time Frame: approximately 15 minutes
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Nicotine Lozenge Prior to Cue Exposure | Placebo Lozenge Prior to Cue Exposure | Control Condition: Lozenge After Cue Exposure
Number analyzed (Participants) | 46 | 46 | 45
units on a scale | 1.28 (0.39) | 0.96 (0.39) | 1.92 (0.39)
Statistical Analysis 1: Comparison: Nicotine Lozenge Prior to Cue Exposure vs Placebo Lozenge Prior to Cue Exposure vs Control Condition: Lozenge After Cue Exposure; Test type: Superiority; p = 0.18, Mixed Models Analysis — Adjusted for treatment order, session, room sequence

ADVERSE EVENTS:
Arm/Group | Nicotine Lozenge Prior to Cue Exposure | Placebo Lozenge Prior to Cue Exposure | Control Condition: Lozenge After Cue Exposure
Serious Adverse Events (participants affected / at risk) | 0/46 | 0/46 | 0/45
Other Adverse Events (participants affected / at risk) | 0/46 | 0/46 | 0/45

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less